CLINICAL TRIAL: NCT02905435
Title: A Traditional Feasibility Study to Assess the Safety and Effectiveness of the Biodegradable Temporizing Matrix (BTM) in the Treatment of Deep Burn Skin Injuries.
Brief Title: Assessment of Safety and Effectiveness of Biodegradable Temporizing Matrix in the Treatment of Deep Burn Skin Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PolyNovo Biomaterials Pty Ltd. (Industry)
Collaborators: PPD Development, LP (Industry); Department of Health and Human Services (U.S. Federal Agency); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-002
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Burns
Keywords: burns; autografts; humans; biodegradable polyurethane; dermal matrix; synthetic
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biodegradable Temporizing Matrix (Experimental): Biodegradable Temporizing Matrix (BTM)
  Interventions: Device: Biodegradable Temporizing Matrix

INTERVENTIONS:
Device: Biodegradable Temporizing Matrix — The Biodegradable Temporizing Matrix (BTM) (also known as NovoSorb BTM) comprises a completely synthetic, sterile, integrating dermal component (porous biodegradable polyurethane foam) and a temporary epidermal barrier component (a non-biodegradable polyurethane sealing membrane). These layers are adhered with a biodegradable polyurethane bonding layer. BTM will be implanted and fixed into position to close a debrided burn wound. After a period of integration, the sealing membrane is removed and a split skin graft is applied.

SUMMARY:
This is a multi-center, single arm, traditional feasibility study to allow a preliminary assessment of the safety and effectiveness of a new method of treating skin burns using Biodegradable Temporizing Matrix (BTM).

DETAILED DESCRIPTION:
This is a multi-center, single arm, traditional feasibility study to allow a preliminary assessment of the safety and effectiveness of BTM treatment. Patients with 10-70% TBSA burns will have BTM devices implanted in areas with deep partial or full thickness burns to treat at least 5% TBSA.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent (directly or via legal representative) prior to any clinical trial procedures being performed.
* Willing to comply with all study procedures and expects to be available for the duration of the study.
* Male and non-pregnant females ≥ 18 years of age and ≤ 70 years of age.
* Patients with deep partial or full thickness burns (between 10% and 70% inclusive of their TBSA).

Exclusion Criteria:

* Has a known hypersensitivity to polyurethane or silver-containing materials.
* Multiple traumas (significant traumatic injury to a solid organ in addition to skin).
* Presence of a medical condition with a life expectancy of less than 12 months, such as advanced malignancy.
* Presence of a medical condition that might interfere with treatment evaluation; or require a change in therapy including but not limited to, significant immune deficiency, or skin or vascular diseases in the area of the wound.
* Female with known or suspected pregnancy, planned pregnancy, or lactation.
* Has had exposure to any other investigational agent within the last 6 months.
* Has a clinically significant psychiatric illness.
* Has a condition the Investigator believes would interfere with the ability to comply with study instructions, or that might confound the interpretation of the study results or put the subject at undue risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-11-05 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus JD Wagstaff, MBBS, PhD, Principal Investigator — Royal Adelaide Hospital, Adelaide SA 5000, AUSTRALIA
Locations (5):
- United States (5):
  - Arizona Burn Center at Maricopa Medical Center, Phoenix, Arizona
  - University of California Davis Medical Center, Sacramento, California
  - Tampa General Hospital, Tampa, Florida
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — https://polynovo.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only participants (or their legally authorized representatives) who provided written informed consent and who met the eligibility criteria were enrolled and had BTM applied to the study lesions. Participants (or their legally authorized representatives) who provided informed consent but who did not meet the eligibility criteria were excluded and did not have BTM applied.
Groups:
- Biodegradable Temporizing Matrix: Biodegradable Temporizing Matrix (BTM)
  Biodegradable Temporizing Matrix: The Biodegradable Temporizing Matrix (BTM) (also known as BTM Dressing) comprises a completely synthetic, sterile, integrating dermal component (porous biodegradable polyurethane foam) and a temporary epidermal barrier component (a non-biodegradable polyurethane sealing membrane). These layers are adhered with a biodegradable polyurethane bonding layer. BTM will be implanted and fixed into position to close a debrided burn wound. After a period of integration, the sealing membrane is removed and a split skin graft is applied.
Period: Overall Study
Arm/Group | Biodegradable Temporizing Matrix
Started | 14
Completed | 7
Not Completed | 7
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Biodegradable Temporizing Matrix
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (15.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 14
Height [Mean (Standard Deviation); unit: centimetres] | 174.1 (10.4)
Weight [Mean (Standard Deviation); unit: kilograms] | 93.0 (26.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/metre^2] | 30.8 (8.3)
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick skin type describes a way to classify the skin by its reaction to exposure to sunlight. Skin types are based on questions posed to study participants that reflect the color of their eyes, hair, skin and the response of the skin when exposed to the sun. Participants are categorized in a range from Type I to Type VI, with Type I corresponding to light skin and Type VI to dark skin.
  Participants
    Type I | 0
    Type II | 2
    Type III | 7
    Type IV | 1
    Type V | 1
    Unknown | 3
Burn Etiology [Count of Participants; unit: Participants]
  Thermal | 13
  Other (Contact) | 1
% Total Body Surface Area (TBSA) affected by deep dermal/full thickness burn injury [Mean (Full Range); unit: Percentage of total body surface area] | 45.1 [10 to 70]

OUTCOME MEASURES:

1. Primary Outcome: BTM 'Take' Rate
Description: Percentage of total body surface area (%TBSA) of BTM that has adhered at time of skin grafting, divided by the %TBSA treated with BTM, then multiplied by 100 to express as a percentage. Calculated per study lesion and averaged per participant.
Time Frame: At time of application of split skin graft (SSG) (typically 28-35 days after application of BTM, Day 0)
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of BTM take per subject
Groups:
- Biodegradable Temporizing Matrix (BTM): The Biodegradable Temporizing Matrix (BTM) (also known as NovoSorb BTM) comprises a completely synthetic, sterile, integrating dermal component (porous biodegradable polyurethane foam) and a temporary epidermal barrier component (a non-biodegradable polyurethane sealing membrane). These layers are adhered with a biodegradable polyurethane bonding layer. BTM will be implanted and fixed into position to close a debrided burn wound. After a period of integration, the sealing membrane is removed and a split skin graft is applied.
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 12
percentage of BTM take per subject | 95.22 (7.175)

2. Primary Outcome: SSG 'Take' Rate Over BTM
Description: The amount (calculated as a percentage) of split skin graft (SSG) that 'takes' expressed as a proportion of SSG applied at 7-10 days after application of SSG. Calculated per study lesion and averaged for each participant.
Time Frame: 7-10 days after application of SSG
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of SSG take per subject
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 11
percentage of SSG take per subject | 97.53 (7.501)

3. Primary Outcome: Adverse Events
Description: Number and type of Adverse Events occurring after BTM implantation
Time Frame: All timepoints until 12 months after application of SSG
Population: Intention to treat
Measure: Number; unit: adverse events
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 14
adverse events
  Any adverse event | 340
  Any adverse event leading to treatment discontinuation | 3
  Any NCI CTCAE Grade 3 or higher adverse event | 8
  Any device-related adverse event | 3
  Any serious adverse event (SAE) | 6
  Any adverse event leading to death | 2
  Any unanticipated adverse device effect (UADE) adverse event | 0

4. Secondary Outcome: Infection
Description: Incidence of infections in BTM-treated areas, and the success of treatment of local infections with BTM in place. Results will be combined and expressed as local infection rate and response rate to treatment.
Time Frame: From day of application (Day 0) until 12 months after SSG.
Measure: Count of Units; unit: Wounds treated with BTM
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 14
Number analyzed (Wounds treated with BTM) | 33
Wounds treated with BTM
  Not infected | 21
  Infected | 12
  Infected - study device retained | 7
  Infected - study device partially removed | 2
  Infected - study device totally removed | 3

5. Secondary Outcome: Wound Closure - Anterior Torso
Description: Clinical assessment of wound closure expressed as a percentage, per anatomical region
Time Frame: 1, 2, 3, 6, 12 months after application of SSG
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: % wound closure
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 5
Number analyzed (Wounds treated with BTM) | 5
% wound closure
  1 month after SSG | 99.8 (0.45)
  2 months after SSG: number analyzed (Wounds treated with BTM) | 4
  2 months after SSG | 99.8 (0.5)
  3 months after SSG: number analyzed (Wounds treated with BTM) | 4
  3 months after SSG | 99.8 (0.5)
  6 months after SSG: number analyzed (Wounds treated with BTM) | 4
  6 months after SSG | 100.0 (0)
  12 months after SSG: number analyzed (Wounds treated with BTM) | 3
  12 months after SSG | 100 (0)

6. Secondary Outcome: Wound Closure - Left Lower Limb
Description: Clinical assessment of wound closure expressed as a percentage, per anatomical region
Time Frame: 1, 2, 3, 6, 12 months after application of SSG
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: % wound closure
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 5
Number analyzed (Wounds treated with BTM) | 5
% wound closure
  1 month after SSG: number analyzed (Wounds treated with BTM) | 4
  1 month after SSG | 95.8 (4.27)
  2 months after SSG: number analyzed (Wounds treated with BTM) | 4
  2 months after SSG | 95.8 (4.27)
  3 months after SSG | 100 (0)
  6 months after SSG: number analyzed (Wounds treated with BTM) | 4
  6 months after SSG | 100 (0)
  12 months after SSG: number analyzed (Wounds treated with BTM) | 3
  12 months after SSG | 100 (0)

7. Secondary Outcome: Wound Closure - Left Upper Limb
Description: Clinical assessment of wound closure expressed as a percentage, per anatomical region
Time Frame: 1, 2, 3, 6, 12 months after application of SSG
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: % wound closure
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 3
Number analyzed (Wounds treated with BTM) | 3
% wound closure
  1 month after SSG | 100.0 (0)
  2 months after SSG | 100.0 (0)
  3 months after SSG | 100.0 (0)
  6 months after SSG | 100.0 (0)
  12 months after SSG | 100.0 (0)

8. Secondary Outcome: Wound Closure - Posterior Torso
Description: Clinical assessment of wound closure expressed as a percentage, per anatomical region
Time Frame: 1, 2, 3, 6, 12 months after application of SSG
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: % wound closure
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 6
Number analyzed (Wounds treated with BTM) | 6
% wound closure
  1 month after SSG: number analyzed (Wounds treated with BTM) | 4
  1 month after SSG | 94.8 (9.84)
  2 months after SSG: number analyzed (Wounds treated with BTM) | 5
  2 months after SSG | 95.8 (8.84)
  3 months after SSG | 100.0 (0)
  6 months after SSG | 100.0 (0)
  12 months after SSG: number analyzed (Wounds treated with BTM) | 5
  12 months after SSG | 99.6 (0.89)

9. Secondary Outcome: Wound Closure - Right Lower Limb
Description: Clinical assessment of wound closure expressed as a percentage, per anatomical region
Time Frame: 1, 2, 3, 6, 12 months after application of SSG
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: % wound closure
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 5
Number analyzed (Wounds treated with BTM) | 5
% wound closure
  1 month after SSG: number analyzed (Wounds treated with BTM) | 4
  1 month after SSG | 96.0 (4.52)
  2 months after SSG: number analyzed (Wounds treated with BTM) | 4
  2 months after SSG | 96.3 (4.79)
  3 months after SSG | 99.8 (0.45)
  6 months after SSG: number analyzed (Wounds treated with BTM) | 4
  6 months after SSG | 99.8 (0.50)
  12 months after SSG: number analyzed (Wounds treated with BTM) | 3
  12 months after SSG | 99.7 (0.58)

10. Secondary Outcome: Ease of Use: "BTM is Easy to Use"
Description: Operator ease of use as determined by physician survey, scored on a 1 to 5 scale, where 1 = strongly agree and 5 = strongly disagree.
  A higher score means a worse outcome.
Time Frame: At time of application of SSG (typically 28-35 days after application of BTM, Day 0)
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 14
Number analyzed (Wounds treated with BTM) | 33
score on a scale
  Site 1: number analyzed (Participants) | 1
  Site 1: number analyzed (Wounds treated with BTM) | 2
  Site 1 | 2.0 (0)
  Site 3: number analyzed (Participants) | 1
  Site 3: number analyzed (Wounds treated with BTM) | 2
  Site 3 | 1.0 (0)
  Site 4: number analyzed (Participants) | 8
  Site 4: number analyzed (Wounds treated with BTM) | 18
  Site 4 | 1.7 (0.69)
  Site 5: number analyzed (Participants) | 3
  Site 5: number analyzed (Wounds treated with BTM) | 8
  Site 5 | 1.0 (0)

11. Secondary Outcome: Ease of Use: "BTM is Easy to Apply"
Description: as for outcome 10
Time Frame: At time of application of SSG (typically 28-35 days after application of BTM, Day 0)
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 14
Number analyzed (Wounds treated with BTM) | 33
score on a scale
  Site 1: number analyzed (Participants) | 1
  Site 1: number analyzed (Wounds treated with BTM) | 2
  Site 1 | 2.0 (0)
  Site 3: number analyzed (Participants) | 1
  Site 3: number analyzed (Wounds treated with BTM) | 2
  Site 3 | 1.0 (0)
  Site 4: number analyzed (Participants) | 8
  Site 4: number analyzed (Wounds treated with BTM) | 18
  Site 4 | 1.8 (0.94)
  Site 5: number analyzed (Participants) | 3
  Site 5: number analyzed (Wounds treated with BTM) | 8
  Site 5 | 1.0 (0)

12. Secondary Outcome: Ease of Use: "BTM is Easy to Delaminate"
Description: as for outcome 10
Time Frame: At time of application of SSG (typically 28-35 days after application of BTM, Day 0)
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 14
Number analyzed (Wounds treated with BTM) | 33
score on a scale
  Site 1: number analyzed (Participants) | 1
  Site 1: number analyzed (Wounds treated with BTM) | 2
  Site 1 | 1.0 (0)
  Site 3: number analyzed (Participants) | 1
  Site 3: number analyzed (Wounds treated with BTM) | 2
  Site 3 | 1.0 (0)
  Site 4: number analyzed (Participants) | 7
  Site 4: number analyzed (Wounds treated with BTM) | 16
  Site 4 | 1.2 (0.40)
  Site 5: number analyzed (Participants) | 3
  Site 5: number analyzed (Wounds treated with BTM) | 8
  Site 5 | 1.0 (0)

13. Secondary Outcome: Ease of Use: "BTM is a Product I Would Use for Other Burn Patients"
Description: as for outcome 10
Time Frame: At time of application of SSG (typically 28-35 days after application of BTM, Day 0)
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 14
Number analyzed (Wounds treated with BTM) | 33
score on a scale
  Site 1: number analyzed (Participants) | 1
  Site 1: number analyzed (Wounds treated with BTM) | 2
  Site 1 | 2.0 (0)
  Site 3: number analyzed (Participants) | 1
  Site 3: number analyzed (Wounds treated with BTM) | 2
  Site 3 | 1.0 (0)
  Site 4: number analyzed (Participants) | 7
  Site 4: number analyzed (Wounds treated with BTM) | 16
  Site 4 | 1.3 (0.60)
  Site 5: number analyzed (Participants) | 3
  Site 5: number analyzed (Wounds treated with BTM) | 8
  Site 5 | 1.0 (0)

14. Secondary Outcome: Joint Contracture
Description: Joint contracture after treatment, assessed by Joint Contracture Severity Scale. Joint Contracture Severity Scale is assessed per anatomical joint and assigned a value from 1 to 3, where 1 = Mild, 2 = Moderate, 3 = Severe.
  Results summarized as the number of participants who had at least one joint assessed with a joint contracture of each severity grade. Where more than one joint motion was affected (e.g. knee flexion, knee extension, etc.), the motion with the most severe contracture at a specific timepoint was reported in the summary results.
Time Frame: 1, 2, 3, 6, 12 months after application of BTM
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 14
Participants
  1 month after SSG: number analyzed (Participants) | 4
  1 month after SSG: 1, Mild | 2
  1 month after SSG: 2, Moderate | 1
  1 month after SSG: 3, Severe | 1
  2 months after SSG: number analyzed (Participants) | 4
  2 months after SSG: 1, Mild | 2
  2 months after SSG: 2, Moderate | 1
  2 months after SSG: 3, Severe | 1
  3 months after SSG: number analyzed (Participants) | 3
  3 months after SSG: 1, Mild | 2
  3 months after SSG: 2, Moderate | 1
  3 months after SSG: 3, Severe | 0
  6 months after SSG: number analyzed (Participants) | 4
  6 months after SSG: 1, Mild | 3
  6 months after SSG: 2, Moderate | 1
  6 months after SSG: 3, Severe | 0
  12 months after SSG: number analyzed (Participants) | 4
  12 months after SSG: 1, Mild | 3
  12 months after SSG: 2, Moderate | 1
  12 months after SSG: 3, Severe | 0

15. Secondary Outcome: Scar Severity
Description: Scar appearance/quality assessed by the Modified Vancouver Scar Scale (mVSS), which includes 4 individual sub-scale scores of Pigmentation, Vascularity, Pliability, and Height (mm) of burn lesion and a Total of the individual sub-scale scores.
  Pigmentation: 0=Normal color, 1=Hypopigmentation, 2=Hyperpigmentation, 3=Combination/Mixed Vascularity: 0=Normal, 1=Pink, 2=Red, 3=Purple. Pliability: 0=Normal, 1=Supple, 2=Yielding, 3=Firm, 4=Banding, 5=Contracture. Height (mm): 0=Normal (flat), 1='<2', 2='>2 and <5', 3='>=5' Total: Sum of individual mVSS scores. Minimum total value = 0. Maximum total value = 14.
  Higher scores mean a worse outcome.
Time Frame: 1, 2, 3, 6 and 12 months after application of SSG
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: Total score on a scale
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix (BTM)
Number analyzed (Participants) | 14
Number analyzed (Wounds treated with BTM) | 33
Total score on a scale
  1 month after SSG: number analyzed (Participants) | 10
  1 month after SSG: number analyzed (Wounds treated with BTM) | 20
  1 month after SSG | 7.3 (2.7)
  2 months after SSG: number analyzed (Participants) | 9
  2 months after SSG: number analyzed (Wounds treated with BTM) | 22
  2 months after SSG | 7.7 (1.78)
  3 months after SSG: number analyzed (Participants) | 10
  3 months after SSG: number analyzed (Wounds treated with BTM) | 23
  3 months after SSG | 6.7 (1.61)
  6 months after SSG: number analyzed (Participants) | 9
  6 months after SSG: number analyzed (Wounds treated with BTM) | 23
  6 months after SSG | 6.4 (2.76)
  12 months after SSG: number analyzed (Participants) | 7
  12 months after SSG: number analyzed (Wounds treated with BTM) | 17
  12 months after SSG | 4.5 (2.24)

16. Secondary Outcome: Skin Itch
Description: Pruritus incidence and severity assessed by Numerical Rating Scale from 0 to 10, where 0 = no itch and 10 = worst itch imaginable.
  Higher scores mean a worse outcome.
Time Frame: At 1, 2, 3, 6, 12 months after application of SSG
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Wounds treated with BTM
Arm/Group | Biodegradable Temporizing Matrix
Number analyzed (Participants) | 14
Number analyzed (Wounds treated with BTM) | 33
score on a scale
  1 month after SSG: number analyzed (Participants) | 10
  1 month after SSG: number analyzed (Wounds treated with BTM) | 20
  1 month after SSG | 2.8 (4.05)
  2 months after SSG: number analyzed (Participants) | 9
  2 months after SSG: number analyzed (Wounds treated with BTM) | 20
  2 months after SSG | 2.4 (3.52)
  3 months after SSG: number analyzed (Participants) | 10
  3 months after SSG: number analyzed (Wounds treated with BTM) | 23
  3 months after SSG | 3.3 (3.35)
  6 months after SSG: number analyzed (Participants) | 9
  6 months after SSG: number analyzed (Wounds treated with BTM) | 21
  6 months after SSG | 3.7 (3.35)
  12 months after SSG: number analyzed (Participants) | 7
  12 months after SSG: number analyzed (Wounds treated with BTM) | 17
  12 months after SSG | 4.4 (4.18)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the study period of up to 12 months after application of the split-thickness skin graft.
Arm/Group | Biodegradable Temporizing Matrix
All-Cause Mortality (participants affected / at risk) | 2/14
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biodegradable Temporizing Matrix (N=14)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) — Infected pseudoaneurysm of right femoral artery
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 2 (2) — Loss of airway
Fusarium infection (Infections and infestations) | 1 (1) — Fusarium skin infection
Sepsis (Infections and infestations) | 1 (1) — Sepsis
Cellulitis infection right lower limb (Infections and infestations) | 1 (1) — Cellulitis infection right lower limb
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) — Intraperitoneal bleeding
Arterial rupture (Vascular disorders) | 1 (1) — Right femoral artery blowout, s/p right femoral artery patch angioplasty with autogenous vein and sartorius muscle flap
Joint contracture on left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Joint contracture
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biodegradable Temporizing Matrix (N=14)
Abdominal distention (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8)
Diarrhoae (Gastrointestinal disorders) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal dilatation (Gastrointestinal disorders) | 1 (1)
Megacolon (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (9)
Oral pain (Gastrointestinal disorders) | 1 (1)
Peritoneal haematoma (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Abscess limb (Infections and infestations) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 2 (2)
Clostridium infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Enterobacter infection (Infections and infestations) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1)
Escherichia infection (Infections and infestations) | 3 (3)
Fungal skin infection (Infections and infestations) | 2 (2)
Haemophilus infection (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1)
Pseudomonas infection (Infections and infestations) | 2 (2)
Purulent discharge (Infections and infestations) | 2 (3)
Skin candida (Infections and infestations) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 5 (11)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Systemic candida (Infections and infestations) | 2 (2)
Tinea pedis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 2 (2)
Wound infection pseudomonas (Infections and infestations) | 2 (3)
Wound infection staphylococcal (Infections and infestations) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 3 (6)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Application site haematoma (General disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 4 (4)
Pain (General disorders) | 3 (3)
Physical deconditioning (General disorders) | 3 (3)
Pyrexia (General disorders) | 5 (5)
Acute stress disorder (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 4 (5)
Delirium (Psychiatric disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (8)
Nightmare (Psychiatric disorders) | 4 (4)
Restlessness (Psychiatric disorders) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 (3)
Incision site pruritus (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 1 (1)
Skin scar contracture (Injury, poisoning and procedural complications) | 3 (4)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 7 (10)
Pelvic vein thrombosis (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Aspergillus test positive (Investigations) | 1 (1)
Blood calcium decreased (Investigations) | 1 (2)
Blood glucose decreased (Investigations) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (2)
Blood phosphorus increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 3 (9)
Enterococcus test positive (Investigations) | 1 (1)
Fungal test positive (Investigations) | 2 (4)
Haemoglobin decreased (Investigations) | 1 (8)
Herpes simplex test positive (Investigations) | 1 (1)
Influenza virus test positive (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pseudomonas test positive (Investigations) | 2 (2)
Staphylococcus test positive (Investigations) | 3 (4)
Trichomonal test positive (Investigations) | 1 (1)
Urine output decreased (Investigations) | 3 (5)
Weight decreased (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Extremity contracture (Musculoskeletal and connective tissue disorders) | 3 (6)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelactasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased viscosity of bronchial secretions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Eye movement disorder (Eye disorders) | 1 (1)
Scleral oedema (Eye disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (2)
Peroneal nerve palsy (Nervous system disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cortisol deficiency (Endocrine disorders) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT02905435/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT02905435/SAP_001.pdf